CLINICAL TRIAL: NCT00906633
Title: Seifem Observational Study of Antifungal Combination Therapy In Hematologic Italian Centers
Brief Title: Seifem Surveillance of Antifungal Combination Therapy In Hematologic Italian Centers
Acronym: SEIFEM COMBO
Status: Completed | Type: Observational
Sponsor: University Hospital, Udine, Italy (Other)
Collaborators: Catholic University of the Sacred Heart (Other)
Responsible Party: CANDONI ANNA, UNIVERSITY HOSPITAL, Udine, Italy
Other Study IDs: SEIFEMcombo0509
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2009-05

CONDITIONS: Fungal Infection
Keywords: antifungal therapies
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Outcome of combination antifungal therapy

SUMMARY:
This trial is an observational study about combination antifungal therapy in hematologic patients with proven and probable invasive fungal infections (IFI).

ELIGIBILITY:
Inclusion Criteria:

* Haematologic patients with proven or probable IFI
* Therapy with a combination of antifungal drugs

Exclusion Criteria:

* Haematologic patients with possible IFI

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Haematologic patients with proven or probable invasive fungal infectious
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
safety, efficacy and duration of therapy | one year

CONTACTS AND LOCATIONS:
Overall Officials: ANNA CANDONI, MD, Principal Investigator — University Hospital, Udine, Italy
Locations (1):
- University Hospital, Udine, Udine, Italy

REFERENCES:
- [Derived] Candoni A, Caira M, Cesaro S, Busca A, Giacchino M, Fanci R, Delia M, Nosari A, Bonini A, Cattaneo C, Melillo L, Caramatti C, Milone G, Scime' R, Picardi M, Fanin R, Pagano L; SEIFEM GROUP (Sorveglianza Epidemiologica Infezioni Fungine nelle Emopatie Maligne). Multicentre surveillance study on feasibility, safety and efficacy of antifungal combination therapy for proven or probable invasive fungal diseases in haematological patients: the SEIFEM real-life combo study. Mycoses. 2014 Jun;57(6):342-50. doi: 10.1111/myc.12161. Epub 2013 Dec 23. PMID 24373120